CLINICAL TRIAL: NCT07391683
Title: Prospective, Randomized Open Label Trial of Telemedically Assisted Optimization for Heart Failure Patients Before Cardiac Surgery to Improve Perioperative Outcome
Brief Title: Telemedically Assisted Optimization for Heart Failure Patients Before Cardiac Surgery to Improve Perioperative Outcome
Acronym: PREPARE-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1169/2025
Record Dates: First submitted 2026-01-07; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Patients With Heart Failure Undergoing Cardiac Surgery
Keywords: cardiac surgery; heart failure; Telemedically Assisted optimization program; prehab; Cardiac Surgical Procedures; Perioperative Care; Preoperative Exercise; Remote Patient Monitoring; Telemedicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Masking Description: Blinding is not feasible because the intervention involves overt telemedical monitoring, patient education, and individualized therapeutic adjustments that are readily apparent to both patients and healthcare providers, necessitating an open-label study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm - Standard of care treatment (No Intervention): Receives standard preoperative care until surgery.
- PREPARE-HF (Experimental): Preoperative Heart Failure Optimization and Telemedicine Integration
  Interventions: Other: PREPARE-HF disease management program, which includes:

INTERVENTIONS:
Other: PREPARE-HF disease management program, which includes: — 1. Heart failure education and training
  2. Optimization of guideline-directed medical therapy (GDMT)
  3. Telemedical / telenursing / monitoring and therapy adjustments
  4. Supervised telemedicine-assisted exercise program
  Arms: PREPARE-HF

SUMMARY:
Patients with heart failure undergoing cardiac surgery face a significantly increased perioperative risk, yet no standardized strategy exists to mitigate this risk effectively. Current preoperative management relies on optimization of medical therapy without a structured prehabilitation approach. Given the strong association between eleveated preoperative N-terminal pro-B-type natriuretic peptide levels and postoperative outcomes, patients at increased risk could be identified using this biomarker. Telemedical disease management programs have demonstrated efficacy in outpatient heart failure care, but their role in preoperative optimization remains underexplored. This study aims to assess whether a structured, multidisciplinary, telemedicine-assisted prehabilitation program can reduce perioperative complications, and improve surgical outcomes.

DETAILED DESCRIPTION:
Patients with heart failure undergoing elective cardiac surgery represent a particularly vulnerable population with a substantially increased risk of perioperative morbidity and mortality. Despite advances in surgical techniques and perioperative care, adverse outcomes such as early postoperative mortality, need for extracorporeal membrane oxygenation (ECMO)need for temporary renal replacement therapy, , and prolonged intensive care unit (ICU) stay,remain frequent in this high-risk group. Current perioperative management largely relies on outpatient treating physicians to optimize guideline-directed medical therapy (GDMT) without a structured, standardized strategy for preoperative optimization or "prehabilitation" tailored to heart failure patients. A key issue for resource intensive optimization programs is the need for good patient selection to identify high-risk patients. N-terminal pro-B-type natriuretic peptide (NT-proBNP) is a well-established biomarker reflecting cardiac wall stress and neurohormonal activation. Elevated NT-proBNP levels are independently associated with adverse perioperative and long-term outcomes in patients undergoing both non-cardiac and cardiac surgery. Retrospective data from large surgical cohorts, including analyses from our center, have demonstrated that high preoperative NT-proBNP levels are linked to increased ICU length of stay, higher rates of renal replacement therapy and ECMO use, as well as increased short- and long-term mortality. Importantly, an improvement in measured NT-proBNP levels,reflecting improved heart failure status, were associated with significantly better perioperative outcomes, suggesting that NT-proBNP is not only a risk marker but also identifies potentially optimizable patients. Telemedical disease management programs have proven effective in outpatient heart failure care by improving adherence to GDMT, enabling early detection of clinical deterioration, and reducing hospitalizations. However, the application of such structured telemedicine-assisted interventions in the preoperative setting of cardiac surgery has not been systematically evaluated. The perioperative period offers a unique therapeutic window in which optimization of volume status, neurohormonal blockade, functional capacity, and patient education may translate into improved surgical readiness and outcomes. The PREPARE-HF project was designed to address this unmet clinical need by evaluating a multidisciplinary, telemedicine-assisted preoperative optimization program for high-risk heart failure patients scheduled for elective cardiac surgery. The intervention integrates structured heart failure education, optimization of guideline-directed medical therapy, continuous telemonitoring, supervised exercise training, and psychological support, with the aim of improving perioperative complications compared with standard of care. PREPARE-HF is conducted as a prospective, randomized, open-label ontrolled clinical trial in which 162 patients with elevated NT-proBNP levels (≥1500 ng/L) are randomized in a 1:1 ratio to either the intervention program or standard preoperative care, with stratification according to surgical procedure type. The primary endpoint is a hierarchical composite outcome assessed using the Finkelstein-Schoenfeld win ratio methodology, incorporating all-cause mortality, need for extracorporeal membrane oxygenation, requirement for renal replacement therapy, and length of intensive care unit stay within 30 days after surgery. Secondary endpoints include safety endpoints, preoperative events, perioperative complications, short- and long-term mortality, functional capacity, quality of life, biomarker dynamics, and adherence to guideline-directed heart failure therapy, enabling a comprehensive assessment of the intervention's impact on perioperative and long-term outcomes in this vulnerable patient population.

ELIGIBILITY:
Inclusion Criteria:

* Indication for elective cardiac surgery in the Heart team
* NTproBNP ≥ 1500 ng/L
* ≥ 18 years willing to participate in trial
* Written informed consent

Exclusion Criteria:

* Neuropsychiatric disorders / illnesses (e.g. drug addiction, alcohol abuse) that do not allow adherent participation in the study
* No sufficient ability to measure and transfer data or existing support in the social environment
* no sufficient ability to communicate (language skills, eyesight, hearing)
* Pregnancy
* Chronic kidney disease requiring dialysis
* Planed procedure: heart transplantation (HTX), implant of left ventricular mechanical assist devices (L-VAD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2034-01-01 (Estimated)

PRIMARY OUTCOMES:
Hierachical Endpoint Perioperative Outcome: 30-day mortality | assessed from randomization through 30 days post-surgery,
  All-cause mortality from randomization to 30 days post-surgery
Hierachical Endpoint Perioperative Outcome: ECMO | assessed from surgery until 30 days post-surgery
  Requirement for extracorporeal membrane oxygenation (ECMO) within 30 days post-surgery
Hierachical Endpoint Perioperative Outcome: hemodialysis or ultrafiltration | assessed from surgery until 30 days post-surgery
  Need for hemodialysis or ultrafiltration within 30 days post-surgery
Hierachical Endpoint Perioperative Outcome: stay on ICU | assessed from surgery until 30 days post-surgery.
  Length of stay in the intensive care unit (ICU) within 30 days post-surgery

SECONDARY OUTCOMES:
Preoperative adverse events: death | will be assessed on day prior to surgery
  Death prior to surgery
Preoperative adverse events: hospitalization | will be assessed on day prior to surgery
  Cardiovascular related hospitalization prior to surgery
Preoperative adverse events: urgent surgery necessary | will be assessed on day prior to surgery
  Urgent cardiac surgery necessary before scheduled surgery date
Perioperative outcome: 30-day mortality | will be assessed on day 30 after surgery
  30-day mortality after surgery
Perioperative outcome: ECMO | will be assessed on day 30 after surgery
  Need for extracorporeal membrane oxygenation (ECMO) within 30 days post-surgery
Perioperative outcome: hemodialysis or ultrafiltration | will be assessed on day 30 after surgery
  Need for hemodialysis or ultrafiltration within 30 days post- surgery
Perioperative outcome: days on ICU | will be assessed on day 30 after surgery
  Duration of stay (days) on intensive care unit within 30 days post-surgery
Preoperative risk assessment | assessed at randomization and on day before surgery
  Change in EuroSCORE II (estimated 30-day mortality, %) from randomization to the pre-operative day.
Quality of guideline-directed heart failure medical therapy (GDMT) | assessed at randomization an on day prior to surgery
  It examines which recommended drug classes patients receive and whether these therapies are prescribed according to current clinical guidelines. In addition, the analysis measures the dosage of each medication and determines the extent to which the prescribed dose corresponds to the percentage of the target dose recommended by the guidelines.
5-year mortality | will be assessed within the 5-years after surgery
  5-year mortality after surgery
EQ-5D-5L | from randomization to postoperative visit at 5 years post-surgery
  Difference in EQ-5D-5L index score (a standardized measure of health-related quality of life developed by the EuroQol Group; range -0.594 to 1.000, with higher scores indicating better health status, 1.000 representing full health, 0 equivalent to death, and negative values indicating health states perceived as worse than death) from baseline to each time point.
EHFScB | from randomization to postoperative visit at 5 years post-surgery
  Difference in the European Heart Failure Self-care Behaviour Scale (EHFScB; a standardized measure of heart failure-related self-care behaviour; score range 0-100, with lower scores indicating better self-care behaviour and higher scores indicating poorer self-care) from baseline to each time point.
GAD-7 | assessed at randomization and on day before surgery
  Difference in the Generalized Anxiety Disorder 7-item scale (GAD-7; a standardized measure of anxiety severity; score range 0-21, with higher scores indicating greater anxiety severity: 0-4 minimal, 5-9 mild, 10-14 moderate, and 15-21 severe anxiety) from baseline to each time point.
6-minute walk test | assessed at randomization and on day prior to surgery
  Changes in 6-minute walk test from baseline to preoperative visit will be evaluated.
1-minute sit to stand test | assessed at randomization and on day prior to surgery
  Changes in 1-minute sit to stand test from baseline to preoperative visit will be evaluated.
NT-proBNP | assessed at randomization and on day prior to surgery
  Changes in NT-proBNP values from baseline to preoperative visit will be evaluated.
Kidney function | assessed at randomization and on day prior to surgery
  Changes in creatinine levels and eGFR from baseline to preoperative visit will be evaluated.
APACHE II Score | daily from the day of surgery until 30 days after surgery, on each day the patient is in the intensive care unit
  Difference in the Acute Physiology and Chronic Health Evaluation II score (APACHE II; a widely used severity-of-disease classification system for critically ill patients; score range 0-71, with higher scores indicating greater disease severity and higher predicted mortality) assessed daily throughout the intensive care unit stay.
NYHA stage | from randomization to postoperative visit at 5 years post-surgery
  Change in New York Heart Association (NYHA) functional class (a clinician-assessed measure of heart failure symptom severity; classes I-IV, with higher classes indicating greater functional limitation) from baseline to each time point.
red blood concentrates | assessed from surgery until 30 days post-surgery
  The necessity for red blood cell concentrates during surgery and within the first 30 days after surgery will be evaluated.
Smoking status | from randomization to postoperative visit at 5 years post-surgery
  Changes in number of smokers from baseline from each time point.
ECHO | assessed at randomization and on day prior to surgery
  Changes in echocardiographic parameters (LV-EF; TAPSE; Severity of valvular heart disease) from baseline to preoperative visit will be evaluated.

OTHER OUTCOMES:
Safety endpoint: Hyperkalemia | from randomization to day prior to surgery
  Hyperkalemia (>6mmol/l) will be assessed as a safety endpoint throughout the PREPARE-HF program.
Safety endpoint: Acute kidney injury | from randomization to day prior to surgery
  Acute kidney injury (>= AKIN 2) will be assessed as a safety endpoint throughout the PREPARE-HF program.
Safety endpoint: Syncope | from randomization to day prior to surgery
  Syncope due to hypotension or bradycardia will be assessed as a safety endpoint throughout the PREPARE-HF program.
Safety endpoint: hospitalization | from randomization to day prior to surgery
  Unplanned hospitalization not due to heart failure or cardiac surgery will be assessed as a safety endpoint throughout the PREPARE-HF program.
Safety endpoint: New permanent contraindication to surgery | from randomization to day prior to surgery
  New permanent contraindication to surgery will be assessed as a safety endpoint throughout the PREPARE-HF program.
Safety endpoint: No need for cardiac surgery | from randomization to day prior to surgery
  No need for cardiac surgery will be assessed as a safety endpoint throughout the PREPARE-HF program.

CONTACTS AND LOCATIONS:
Overall Officials: Can Gollmann-Tepeköylü, Prof., Principal Investigator — Medical University of Innsbruck - Department of cardiac surgery; Gerhard Pölzl, Prof., Principal Investigator — Medical University of Innsbruck - Department of cardiology

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: following publication of primary and secondary results
Access Criteria: Data will be shared upon reasonable request.